CLINICAL TRIAL: NCT02573805
Title: the Evaluation of Diagnostic Value of Rigiscan Test (Nocturnal Penile Tumescence and Rigidity, NPTR) in Chinese Males
Brief Title: the Diagnostic Value of Rigiscan Test (Nocturnal Penile Tumescence and Rigidity, NPTR) in Chinese Males
Acronym: NPTR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Leilei Zhu, doctor leilei zhu, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: NPTR in 2015-09-24
Record Dates: First submitted 2015-10-09; First posted 2015-10-12 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Erectile Dysfunction
Keywords: nocturnal penile tumescence and rigidity; erectile dysfunction; Chinese males
MeSH Terms: conditions — Erectile Dysfunction; Muscle Rigidity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: None Retained — Rigiscan parameters analyzed by Rigiscan plus software
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- erectile dysfunction group: International Index of Erectile Function (IIEF-5) questionnaire≥22 Rigiscan test are performed for two nights
  Interventions: Device: Rigiscan test
- control group: International Index of Erectile Function (IIEF-5) questionnaire<22 Rigiscan test are performed for two nights
  Interventions: Device: Rigiscan test

INTERVENTIONS:
Device: Rigiscan test — Rigiscan tests are performed in enrolled subjects for consecutive two nights.

SUMMARY:
The purpose of this study is to evaluate the diagnostic value of Rigiscan (nocturnal penile tumescence and rigidity, NPTR ) test in erectile dysfunction of Chinese males.

DETAILED DESCRIPTION:
The Rigiscan test is used to evaluate the NPTR parameters. The "normal" NPTR parameter is provided by the Rigiscan manufacturer based on a clinical study on 500 American males. Original studies of NPTR parameters on Chinese males are warranted. On the other hand, during the past decades, several new NPTR parameters have been developed, like tip TAU (tip tumescence activity units), tip RAU (tip rigidity activity units), base TAU (base tumescence activity units), base RAU (base rigidity activity units), but their diagnostic values have been less evaluated. Basd on the these background, we determined to observe the clinical manifestation of these new parameters and to establish the "normal criteria" of NPTR parameters in Chinese males. This could be clinically beneficial in the differential diagnosis of organic and psychological erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. patients in a stable and heterosexual partnership with a fixed sexual partner for more than 6 months;
2. age≥20 year;
3. complete the validated International Index of Erectile Function (IIEF-5) questionnaire.

Exclusion Criteria:

1. advanced age (≥65);
2. pelvic trauma
3. thyroid diseases
4. metabolic diseases
5. hypogonadism and other hormonal disorders
6. sleep disorders
7. penile deformities
8. taking drugs that may interfere with erectile function.

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chinese males ≥20 years
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-08 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Previous Rigiscan parameters analyzed by Rigiscan plus software | within 2 days after the Rigiscan test
  number of erectile events (per night), Duration of tip erections≥60% (min),duration of base erections ≥ 60% (min)

SECONDARY OUTCOMES:
newly developed Rigiscan parameters analyzed by Rigiscan plus software | within 2 days after the Rigiscan test
  RAU tip, TAU tip, RAU base, TAU base, average tip tumescence (cm), average base tumescence(cm), average event rigidity of tip (%),aveage event rigidity of base (%)

CONTACTS AND LOCATIONS:
Overall Officials: l zhu, doctor, Principal Investigator — Drum tower Hospital, school of Medicine, Nanjing University
Locations (1):
- Yutian Dai, Nanjing, Jiangsu, China